CLINICAL TRIAL: NCT04999410
Title: Programming Interval Training Based on the HIIT Classification System on Time-Trial Performance v2
Brief Title: Virtual Programming Interval Training for TT Performance
Acronym: VPHIIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scott G. Thomas (Other)
Collaborators: TrainerRoad (see TrainerRoad.com) (Unknown)
Responsible Party: Sponsor-Investigator, Scott G. Thomas, Professor, University of Toronto
Organization: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: VirtualHIITProgramming01
Record Dates: First submitted 2020-11-29; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Apparently Healthy Adults Cycling Performance
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of four training intervention groups.
  Before to after changes will be contrasted.
Who Masked: Care Provider, Investigator
Masking Description: Employ software to monitor intervention and outcomes. Intervention groups will be coded and the investigators will not be aware of intervention group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Long-HITT (Experimental): Long work bout durations (4 minutes) on cycle ergometers or home trainers
  Interventions: Behavioral: High Intensity Interval Training
- Medium HIIT-L (Active Comparator): Medium duration work bouts (2 minutes) with intensity matched to the Long-HITT intensity
  Interventions: Behavioral: High Intensity Interval Training
- Medium HIIT-H (Active Comparator): Medium duration work bouts (2 minutes) with intensity at 30% of the difference between Wmax and mean TT power outputs
  Interventions: Behavioral: High Intensity Interval Training
- Short HIIT (Active Comparator): Short duration work bouts (30 seconds) with intensity at 50% of the difference between Wmax and mean TT power outputs
  Interventions: Behavioral: High Intensity Interval Training

INTERVENTIONS:
Behavioral: High Intensity Interval Training — Interventions will contrast alternative training protocols

SUMMARY:
High Intensity Interval Training (HIIT) studies are required to determine the optimal training protocol to improve time trial(TT) performance. Data collection for this study will be conducted virtually through the use of a software platform (www.trainerroad.com) by people in their homes on cycle ergometers. Investigators will recruit people who are familiar with cycle exercise training and have their own equipment. By using a virtual platform to collect data, investigators will extend our reach to include a much larger and diverse sample of adult men and women up to age 45 years. In addition, the software platform will allow participants to train from the safety of their home, preventing the risk of exposure to COVID19.

OBJECTIVES O1: The primary objective of this study is to determine the influence of interval work-bout duration on TT performance when total mechanical work is matched.

O2: The secondary objective of the study is to determine the influence of work-bout duration on TT performance when work is matched by effort.

HYPOTHESIS H1: long duration bouts of HIIT will lead to greater improvements in performance compared to short duration bouts due to larger total amount of work completed during the interval sessions.

H2: HIIT will lead to equivalent improvements in performance when work is matched by the participant's rating of effort.

DETAILED DESCRIPTION:
Participants will complete a training history and will be characterized with a questionnaire with respect to age, sex and location. Prior to the first testing session, participants will keep a food diary for the day preceeding the testing session to permit replication of diet for other testing weeks. Participants will be provided with a coded TrainerRoad account used to record all testing and training data. Training sessions will be pre-programmed into the TrainerRoad platform. All testing and training will be completed by participants at their residence on their own bicycles with the use of a smart trainer. Participants will complete an incremental exercise test (IET) to determine their maximal power output (Wmax) and two 40-minute Time Trials (TTs). The IET includes a warmup followed by ramp increases in intensity to a voluntary maximum; typically reached after 8 to 12 min.

Testing will be conducted in the 2-weeks prior and the week following the intervention. Once baseline testing is completed, participants will begin the interval training program which will consist of two interval training sessions per week and 2-3 sessions of low-intensity continuous training. There will be assessor blinding since all testing and training will be conducted solely by the participant with guidance from the TrainerRoad software.

MEASUREMENTS Time-Trial Performance The TT test will be performed by each participant on their own bicycle connected to a smart trainer. Following the warmup, participants will complete a 40-minute TT to determine their maximal sustainable power which corresponds to 7-8/10 on the 10 point Borg RPE scale. For the first TT test, participants will set their workload to 65% of the power achieved from the IET. Participants can consume water ad libitum for the duration of the time trial. Heart rate, cadence, mean power output and maximal power output will be recorded using the TrainerRoad platform.

Maximal Power Output (Wmax). The incremental exercise test determines Wmax. The first stage of the assessment will be completed at the same intensity completed during the warmup phase and increased by 12.5 watts every 30-seconds until the participant is unable to maintain a cadence of 70 RPM. All data will be collected using the TrainerRoad platform.

INTERVENTIONS Participants will be randomly allocated to one of four interval training groups via a computer-generated random sequence. Randomization and allocation will be concealed from the investigators. The groups will consist of a long-HIIT, a medium-HIIT matched to long work, a medium-HIIT that is performed at 15% higher intensity (Medium-HIIT-H), and intermittent short-HIIT (Short-HIIT). Each participant will be aware that they will be completing one of four interval exercise programs, however, they will be blinded to the details of the other programs.

Interval Exercise. Participants will perform a 15-minute warm-up. Following the interval session, they will complete a 10-minute cool down. Interval exercise intensity and durations will be provided through the TrainerRoad program.

Long-HIIT will include 4-repetitions of 6-minute work-bouts with 4-minutes of recovery between bouts. The intensity will be set to 15% of the difference between Wmax and the mean power achieved in the 40-minute TT test.

Medium-HIIT will consist of 12-repetitions of 2-minute work-bouts with 2-minutes of recovery. The Medium-HIIT-L group will exercise at the same intensity as the long-HIIT group whereas the Medium-HIIT-H group will perform the interval sessions at 30% of the difference between Wmax and the mean power achieved in the 40-minute TT test. During recovery-bouts, participants cycle at 40% of the work-bout intensity. Short-HIIT will consist of three sets of 16-repetitions of 30-second work-bouts with 15-seconds of active recovery at 50% of the work-intensity with 4-minutes of active recovery.

Low-Intensity Continuous Training (LICT). In addition to the interval training, participants perform at least 3 sessions of low-intensity continuous training (LICT) for 60-minutes to simulate a polarized training model. The intensity for LICT will be set to 40% of the interval training session power. A polarized training model leads to greater improvements in endurance performance when compared to a threshold training or interval training alone.

DATA COLLECTION All participants will be provided with a coded TrainerRoad account to record all testing and training data. Training sessions will be pre-programmed into the TrainerRoad platform. All testing and training will be completed by participants at their residence on their own bicycles with the use of a smart trainer. The TrainerRoad application will record power output, heart rate and cadence for the duration of each exercise session. At the end of each session, participants will record their session rating of perceived exertion on TrainerRoad.

STATISTICAL ANALYSIS Data analysis will be conducted using R and R-Studio. A comparison of the mean of the performance variables will be assessed using a repeated-measures analysis of the variance (ANOVA) to determine differences between the interval protocols. The primary outcome is change in time-trial mean power. Secondary outcomes include change in maximal power output (Wmax), session rating of perceived exertion, time-trial perceived exertion, and adherence. A subgroup analysis will be conducted from baseline data including age, sex, baseline TT performance and Wmax/kg. If there is a significant difference, a post-hoc analysis will be completed using a paired Student's t-test with Bonferroni correction. The level of significance will be set to a p-value of 0.05. Effect size calculations (Cohen's d) with 95% confidence intervals will be used to determine the magnitude of the effect.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 18 and 45 years of age
2. cycling for a minimum of 3 times per week for the previous 6-months.

   Exclusion Criteria:
3. an injury in the previous 6-months preventing them from completing their normal training routine
4. presence of pathology including cardiovascular diseases (heart attack, hypertension), neurological conditions (stroke, etc.) or metabolic conditions (diabetes).

Participants will be asked to confirm their health status when they complete the intake survey.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Time Trial Performance | 1 week before and 1 to 3 days after interventions
  Change in Time required to complete a 40 kilometer simulated cycle ride

SECONDARY OUTCOMES:
Peak Power Output | Before and 1 to 3 days after interventions
  Change in Maximum power output (Watts) achieved on a incremental cycle test

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring High Performance Sport Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No